CLINICAL TRIAL: NCT06650111
Title: Epidemiology, Diagnosis, Medical Care and Prognosis of Tubulointerstitial Nephritis: Results of a Multicenter Retrospective Cohort Study
Acronym: NETI-MULTI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240673
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Nephritis, Interstitial
Keywords: Tubulointerstitial nephritis (TIN)
MeSH Terms: conditions — Nephritis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human native kidney biopsy from a biological collection for patient care, with fixed fragment stored at room temperature and frozen fragment stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients whose biopsy of the care revealed tubulointerstitial nephritis in the foreground and retained as the main cause of renal dysfunction after etiological investigation.
  The biopsies concerned were carried out between 01/01/2010 and 31/12/2019. The clinical follow-up data of the patients from whom the biopsies were taken will be collected until the date of the last follow-up (before 31/12/2021).
  Interventions: Other: Rereading of biopsies; Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Rereading of biopsies — Rereading of biopsies, blinded to the final diagnosis, by a pathologist specializing in nephropathology. This review includes: an optical microscopy study on a fragment fixed with routine staining, an optical microscopy study on a frozen fragment, an immunohistochemical study on a frozen fragment if available.
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file. The clinical data of the care of patients at whom the biopsies belong will be analyzed until the date of the patient's last follow-up (before 12/31/2021).

SUMMARY:
Tubulointerstitial nephritis (TIN), diagnosed on kidney biopsy, represents a common cause of kidney failure. The etiologies are multiple but the diagnosis of the causative disease is sometimes difficult and the treatment is not completely codified.

The research focuses on the characterization of TIN on the etiological, clinical, biological, therapeutic and prognostic levels in order to improve patient care.

For this purpose, kidney biopsies performed for the diagnosis, kept in a biological collection within the biological resource platforms of the Necker-Enfants Malades hospital and the Georges Pompidou hospital will be centrally reviewed, blinded to the final diagnosis.

DETAILED DESCRIPTION:
Tubulointerstitial nephritis (TIN) is defined as a diverse set of renal pathologies caused by a primary lesion of the interstitial compartment, which most often extends to the associated tubular structures. Renal histology establishes the diagnosis by objectifying different types of lesions associated to varying degrees depending on the etiology and clinical course. These lesions are: an interstitial inflammatory infiltrate whose nature is largely dependent on the etiopathogenic mechanisms of the lesion, diffuse or multifocal interstitial fibrosis, tubular epithelial lesions in the form of tubulitis and/or tubular atrophy.

Research focuses on the characterization of TIN on the etiological, clinical, biological, therapeutic and prognostic levels in order to try to improve patient care. For this:

* 1st step: native kidney biopsies performed to establish the diagnosis and kept in a biological collection within the biological resource platforms of the Necker-Enfants Malades hospital and the Georges Pompidou hospital will be centrally reviewed The review will be performed at the Pathology department of Necker hospital, blinded to the final diagnosis for selection of the biopsies that will be included in the study. Included biopsies will be those with tubulointerstitial nephritis retained as the main cause of renal dysfunction after etiological investigation
* 2nd step: collection of clinical and biological data regarding the diagnosis, management and prognosis
* 3rd step: statistical analysis of the data and consolidation of the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who do not object to the use of their medical data and samples for this research
* With a biopsy of the care on native kidney and subject to a biological collection, finding tubulointerstitial nephritis in the foreground and retained as the main cause of renal dysfunction after etiological investigation.
* Signs of histological activity of the NTI objectified during the centralized rereading and defined by:

  * An inflammation of more than 10% of the surface of the entire cortical parenchyma (fibrous and non-fibrous) or a ti score > or = 1 according to the Banff classification
  * AND/OR the presence of at least one granuloma on the biopsy

Exclusion Criteria:

* No access to medical records for data collection, or insufficient clinical data
* Follow-up less than 3 months
* Histological lesions of the tubulointerstitial sector but related to a hematological, urological, genetic etiology or the direct tubular toxicity of a drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with renal dysfunction whose main cause retained after etiological investigation is tubulointerstitial nephritis and treated at the Necker-Enfants Malades hospital or at the Georges Pompidou European hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evolution of glomerular filtration rate and renal survival | Time 0
  Evolution of glomerular filtration rate and renal survival (defined as the persistence of sufficient renal function not requiring the use of a replacement technique) over time and according to etiology.

SECONDARY OUTCOMES:
Significant association between renal prognosis with specific predictive factors | Time 0
  Significant association between renal prognosis, defined by glomerular filtration rate and/or end-stage renal dysfunction with specific predictive factors. Description of Clinical (age, sex, etiology, high blood pressure, diabetes, early extra-renal purification, AKI stage), biological (peak creatinine, hemoglobin, calcemia, proteinuria, hematuria) and histological factors (interstitial infiltrate, tubulitis, presence of granulomas, fibrosis).
Response to corticosteroid therapy | Time 0
  Evolution of glomerular filtration rate and renal survival over time as a function of corticosteroid treatment.
Association between response to corticosteroid therapy and some histological criteria | Time 0
  Association between response to corticosteroid therapy and some histological criteria. Description of histological criteria : interstitial infiltrate, tubulitis, presence of granulomas, fibrosis.
Evaluate the contribution of histological analysis in etiological diagnosis | Time 0
  Performance of pathologist review in establishing blind histological diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Rabant, M.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No